CLINICAL TRIAL: NCT06287593
Title: The Feasibility of Dynamic Liquid Biopsy Monitoring During Neoadjuvant Treatment for EGFR-mutated NSCLC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Weijia Fang, MD, Professor, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NeoLiq
Record Dates: First submitted 2024-02-23; First posted 2024-03-01 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: EGF-R Positive Non-Small Cell Lung Cancer
Keywords: EGFR positive resectable NSCLC; ctDNA

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- group A (Other): For patients with negative ctDNA after 3 weeks of neoadjuvant TKI treatment, radical resection surgery will be performed after continuing TKI treatment for 9-12 weeks.
  Interventions: Other: ctDNA monitoring
- group B (Other): For patients with positive ctDNA after 3 weeks of neoadjuvant TKI treatment, radical resection surgery will be performed after continuing TKI treatment for 9-12 weeks.
  Interventions: Other: ctDNA monitoring
- group C (Other): For patients with positive ctDNA after 3 weeks of neoadjuvant TKI treatment, radical resection surgery will be performed after 3 cycles of TKI plus chemotherapy.
  Interventions: Other: ctDNA monitoring
- group D (Other): For patients with positive ctDNA after 3 weeks of neoadjuvant TKI treatment, radical resection surgery will be performed after 3 cycles of sequential neoadjuvant PD-1 blockades plus chemotherapy.
  Interventions: Other: ctDNA monitoring

INTERVENTIONS:
Other: ctDNA monitoring — Patients will receive ctDNA monitoring before and after 3 weeks of neoadjuvant 3rd TKI treatment and optimize the neoadjuvant treatment plan based on this.

SUMMARY:
This study aimed to assess the value of dynamic ctDNA monitoring in guiding the development of personalized neoadjuvant treatment strategies for EGFR-mutated NSCLC patients.

DETAILED DESCRIPTION:
This study aimed to prospectively enroll approximately 300 resectable stage II-IIIB (T1-4N0-2M0, excluding T4 with invasion of vital structures and bulky or infiltrative N2) NSCLC patients with histologically confirmed EGFR 19del or L858R mutations. Peripheral blood samples will be collected at baseline before neoadjuvant 3rd-generationEGFR TKI therapy, and ctDNA levels will be quantitatively assessed. For patients with positive baseline ctDNA, peripheral blood will be collected again after 3 weeks of neoadjuvant TKI therapy to assess if ctDNA has turned negative, and HRCT will be performed to evaluate the treatment efficiency simultaneously.

In patients with positive baseline ctDNA, for ctDNA-negative patients after 3 weeks of neoadjuvant TKI treatment, radical resection surgery will be performed after continuing TKI treatment for 9-12 weeks (Group A). For ctDNA-positive patients after 3 weeks of neoadjuvant TKI treatment, in combination with imaging changes in the lesions, a multidisciplinary team (MDT) evaluation will be conducted. After discussion between the attending physicians and the patient, the subsequent treatment will either continue TKI treatment for 9-12 weeks (Group B), undergo 3 cycles of TKI plus chemotherapy (Group C), or undergo sequential neoadjuvant immunotherapy plus chemotherapy for 3 cycles (Group D) before radical resection surgery.The study intends to evaluate the correlation between the rate of major pathological response (MPR) and ctDNA levels at 3 weeks after TKI treatment, to compare the difference in pathological response between ctDNA-negative and ctDNA-positive groups after 3 weeks of neoadjuvant TKI treatment and to evaluate the guiding value of dynamic ctDNA monitoring during neoadjuvant therapy for optimizing subsequent treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Patients should voluntarily join this study and sign the informed consent form
2. Patients diagnosed with resectable stage II-IIIB (T1-4N0-2M0, excluding T4 with invasion of vital structures and bulky or infiltrative N2) NSCLC
3. Patients with EGFR 19del or L858R mutations.
4. Age from 18 to 75 years old, both male and female
5. ECOG score 0-1
6. According to the RECIST v1.1 , patients should have at least one measurable lesion
7. For suspicious mediastinal lymph nodes (including pathological enlargement or PET-CT indicating malignancy, etc.), further sampling is required for pathological diagnosis by EUBS, thoracoscopy, or mediastinoscopy
8. According clinical evaluation, the lung function of patients (such as FVC, FEV1, TLC, FRC, DLco, etc.) should be sufficient for pneumonectomy
9. The function of important organs should meet the following requirements: absolute count of neutrophils ≥ 1.5 × 109/L# Platelets

   ≥ 100 × 109/L# Hemoglobin ≥ 90g/L; Serum albumin ≥ 35g/L; Thyroid hormone (TSH) ≤ 1 × ULN# Serum bilirubin ≤ 1.5 × ULN# ALT and AST ≤ 3 × ULN# International standardized ratio (INR) ≤ 1.5 or prothrombin time (PT) ≤ 1.5 × ULN# Serum creatinine ≤ 1.5 × ULN
10. Female patients at childbearing age are required to use contraceptive measures; for male patients whose partners are women at childbearing age, effective methods of contraception should be used during the trial period

Exclusion Criteria:

1. Patients with other primary malignancies within the past 3 years (excluding cured skin basal cell carcinoma and cervical carcinoma in situ)
2. Patients with active hepatitis B/C
3. Patients with any active autoimmune diseases or a history of autoimmune diseases
4. Patients who are using immunosuppressive agents or require systemic hormone therapy
5. Patients with hypertension but without good control even through antihypertensive medication treatment ; patients with clinical symptoms or diseases related to unsatisfying cardiac function
6. Patients with abnormal coagulation function (INR>2.0, PT>16s)
7. Arterial/venous thrombotic events occurred before screening within 6 months
8. Patients with active infection
9. Patients with congenital or acquired immune dysfunction (such as HIV infection)
10. According to the judgment of the researchers, patients have other factors that may affect the results of the research or cause the research to be terminated

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-04-15 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
the rate of major pathological response (MPR) | up to 17 weeks
  the proportion of patients who achieve MRP among those receiving pneumonectomy

SECONDARY OUTCOMES:
the rate of pathological complete response (pCR) | up to 17 weeks
  the proportion of patients who achieve pCR among those receiving pneumonectomy

CONTACTS AND LOCATIONS:
Overall Officials: Weijia Fang, MD, Principal Investigator — The First Affiliated Hospital, Zhejiang University

IPD SHARING:
Plan to Share IPD: No